CLINICAL TRIAL: NCT05405972
Title: Effects of a Behavioral Intervention With Foster Families: A Randomized Controlled Trial
Brief Title: A Behavioral Intervention With Foster Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000382
Record Dates: First submitted 2022-05-05; First posted 2022-06-06 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Family Relationship; Sibling Relations; Behavior, Social
Keywords: Randomized controlled trial; Behavioral Intervention; Sibling; Foster Care
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Intervention Model Description: This study employed a randomized control trial design of a behavioral intervention with foster families caring for a CDFC as well as a permanent child in the home. The intervention tested is self-paced and delivered via technology to include foster families in rural and underserved locations. Behavioral changes of caregivers and children in the home were predicted to improve family functioning and facilitate healing from relationship-based trauma and its associated symptoms. Stratified randomization was used to assign participants into the experimental or control group. Blinding of the two groups to participants was not done (participants knew whether or not they received the video intervention). However, the team blinded the statistical analysis to group with the use of a statistician. Families assigned to the control did have the opportunity to participate in the intervention post-data collection and analysis and outside of the research protocol.
Masking Description: Randomization to group was blinded and done by an independent statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Receiving Intervention (Experimental): The intervention group receives a link each week connecting them to the videos for both parents and children as well as a communicating/connecting activity. The intervention is self-paced over a 4 week period.
  The intervention was titled the Connected Family Series - For Foster Families (CFS-FF) (further referred to as the intervention) and was created/adapted in partnership from the Connected Family Series (CFS) by psychologists at the Karyn Purvis Institute of Childhood Development (KPICD). A letter of support from the KPICD is available in Appendix D. Adaptation was needed as the original intervention was geared toward adoptive families and excluded foster families. This process was done with the original creator (Dr. Jana Hunsley) with members of the research team and fostering community.
  Interventions: Behavioral: The Connected Family Series - For Foster Families
- Control Group (No Intervention): Families in the control group receive no video links during the 4 week period. Families assigned to the control do have the opportunity to participate in the intervention post-data collection and analysis and outside of the research protocol.

INTERVENTIONS:
Behavioral: The Connected Family Series - For Foster Families — A 4-week program involving videos and activities for both the parent and child in the home.
  Arms: Group Receiving Intervention

SUMMARY:
The purpose of this study is to investigate a behavioral intervention with foster families.

DETAILED DESCRIPTION:
Study Aims: This study aims to investigate a technology-delivered family (sibling inclusive) intervention. Focus is on increasing family hardiness and preparation to care for children with disabilities and special needs in foster care. Three aims include: (1) establish the feasibility of the technology-based, family-centered intervention (2) explore in a preliminary manner the effects of the intervention on stress and relational quality outcomes among family member participants, and (3) an exploratory aim to determine feasibility and preliminary efficacy of the intervention on diurnal salivary cortisol levels within the foster family population.

Methods: This study employs a randomized control trial design of a behavioral intervention with both a control and experimental group. The intervention tested was created in partnership and adapted from the Connected Family Series (CFS) by psychologists at the Karyn Purvis Institute of Childhood Development and is called the Connected Family Series - For Foster Families (CFS-FF). Adaptation was needed as the original intervention was geared toward adoptive families and excluded foster families. The CFS-FF also needed content specific to fostering children with special needs. Stress and relational quality outcomes among members will be measured using the concepts of family hardiness, preparedness, and relationship development through a self-report questionnaire which include the Family Hardiness Index (FHI), the Integrating Foster Children (IFC) subscale from the Casey Foster Applicant Inventory (CFAI), and the Sibling Inventory of Behavior (SIB), respectively. Participation in the study spanned three to four months; one month for recruitment and collection of baseline data, one month for the intervention, and one-month post-intervention data collection. Exploratory aim 3 will be achieved by an objective indicator of stress-related biology, saliva diurnal cortisol rhythm, before and after completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. licensed foster families
2. must have at least one permanent child (biological or adopted) living in the home before the foster or newly adopted child entered the home
3. at least one foster or foster-to-adopt child placed in the home
4. all participants other than the foster or foster-to-adopt child must be proficient in English

Exclusion Criteria:

1. Non-English speaking
2. No permanent sibling between the ages of 7 at 17
3. No current foster placement living in the home
4. Designated as a group home
5. Greater than six children living in the home

Ages: 7 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Family Hardiness Index | Before intervention, up to 2 week
  Psychometrically validated self-report tool for family functioning. Unabbreviated scale title: Family Hardiness Index Min Value: 0 Max Value: 60 Higher Score means better/improvement in hardiness

SECONDARY OUTCOMES:
Sibling Inventory of Behavior | Before intervention, up to 2 weeks
  Psychometrically validated self-report tool for sibling relationships. Unabbreviated scale title: Sibling Inventory of Behavior (Positive) Min Value: 15 Max Value: 75 Higher Score means there are more positive outcomes between the siblings
  Unabbreviated scale title: Sibling Inventory of Behavior (Negative) Min Value: 17 Max Value: 85 Higher Score means there are more negative outcomes between the siblings

OTHER OUTCOMES:
Family Hardiness Index | After intervention, up to 3 months
  Psychometrically validated self-report tool for family functioning. Unabbreviated scale title: Family Hardiness Index Min Value: 0 Max Value: 60 Higher Score means better/improvement in hardiness
Sibling Inventory of Behavior | After intervention, up to 3 months
  Psychometrically validated self-report tool for sibling relationships. Unabbreviated scale title: Sibling Inventory of Behavior (Positive) Min Value: 15 Max Value: 75 Higher Score means there are more positive outcomes between the siblings
  Unabbreviated scale title: Sibling Inventory of Behavior (Negative) Min Value: 17 Max Value: 85 Higher Score means there are more negative outcomes between the siblings

CONTACTS AND LOCATIONS:
Overall Officials: Christine Platt, DNP/PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gypen, L., Vanderfaeillie, J., De Maeyer, S., Belenger, L., & Van Holen, F. (2017). Outcomes of children who grew up in foster care: Systematic-review. Children and Youth Services Review, 76, 74-83 — https://doi.org/10.1016/j.childyouth.2017.02.035
- See also: Gypen, L., West, D., Van Holen, F., & Vanderfaeillie, J. (2020). Birth children of foster carers: How do they experience the foster care placement. Child and Youth Services Review 109, 104703 — https://doi.org/10.1016/j.childyouth.2019.104703
- See also: Vanderfaeillie, J., Van Holen, F., Carlier, E., & Fransen, H. (2018b). Breakdown of foster care placements in Flanders: Incidence and associated factors. Eur Child Adolesc Psychiatry, 27(2), 209-220. — https://doi.org/10.1007/s00787-017-1034-7
- See also: Wojciak, A. S., McWey, L. M., & Waid, J. (2018). Sibling relationships of youth in foster care: A predictor of resilience. Children and Youth Services Review, 84, 247-254. — https://doi.org/10.1016/j.childyouth.2017.11.030

DOCUMENTS (3):
  • Study Protocol (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT05405972/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT05405972/SAP_001.pdf
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT05405972/ICF_002.pdf